CLINICAL TRIAL: NCT00298324
Title: A Randomized Double Blinded Placebo-Controlled Phase III Trial Comparing Cyclosporine Plus Steroids With or Without Myfortic as Primary Treatment for Extensive Chronic Graft Versus Host Disease
Brief Title: Myfortic - Treatment for Extensive cGvHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Novartis (Industry)
Responsible Party: Ruzena Uddin, EBMT
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2005-006178-86; EBMT-LE-0601
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Graft vs Host Disease
Keywords: GvHD; graft versus host disease; extensive; myfortic
MeSH Terms: conditions — Graft vs Host Disease | interventions — Mycophenolic Acid; Prednisone; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myfortic (Active Comparator): Patients in this arm will receive Myfortic + Prednisone + Cyclosporine
  Interventions: Drug: Myfortic
- Standard Care/ Placebo (Other): In this arm patients will receive Prednisone + Cyclosporine + Placebo or Prednisone + Cyclosporine
  Interventions: Drug: Prednisone and Cyclosporine

INTERVENTIONS:
Drug: Myfortic — 1440mg twice daily
  Arms: Myfortic
Drug: Prednisone and Cyclosporine — Prednisone and Cyclosporine given according to protocol. The drugs are tapered according to patient response
  Arms: Standard Care/ Placebo

SUMMARY:
The purpose of this study is to determine whether the response to treatment for extensive chronic Graft versus Host Disease (cGvHD)is improved with the addition of myfortic alongside cyclosporine A and prednisone, compared to the reference treatment of cyclosporine A and prednisone alone.

DETAILED DESCRIPTION:
This clinical trial is a European, multi-center, randomized, double blinded placebo-controlled trial comparing CsA+PDN+MPA versus the reference treatment of CsA+PDN alone + placebo, in patients with extensive chronic GvHD. Randomization will be stratified according to:

* Platelet number (low versus high risk)
* Source of transplantable cells (marrow versus PBSC versus cord blood)

Patients not in progression at 6 weeks post randomization (progression defined as primary failure) will be evaluated for remission (complete or partial) at 3, 6, 9, & 12 months post randomization

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60
* Any primary diagnosis requiring treatment by hematopoietic stem cell transplantation
* Recipient of a single allogeneic stem cell transplant (bone marrow or peripheral blood stem cells, or cord blood) minimum 80 days ago
* Received a graft from a related or an unrelated donor
* Conditioning regimen: Myeloablative or non-myeloablative
* Patients suffering a first episode of extensive chronic GvHD, without recurrent disease
* The diagnosis of chronic GvHD requires the following:

  * Distinction from acute GvHD
  * Presence of at least one diagnostic clinical sign of chronic GvHD or presence of at least one distinctive sign confirmed by pertinent biopsy or other relevant diagnostic tests
  * Exclusion of other possible diagnoses
* Receiving a standard prophylaxis regimen for acute GvHD: CsA plus methotrexate, or CSA+MMF for NMA, or a T-cell depleted transplant
* Patient gives written informed consent prior to randomization

Exclusion Criteria:

* Patient age less than 18 years or over 60 years.
* GvHD prophylaxis by tacrolimus plus methotrexate
* Delayed onset acute GvHD following NMA or DLI
* Second allogeneic stem cell transplant
* Not the first episode of chronic GvHD needing systemic immunosuppressive therapy.
* Limited chronic GvHD (Seattle criteria, see Appendix 1)
* Uncontrolled systemic infection which in the opinion of the investigator is associated with an increased risk of the patient's death within 1 week of randomization
* In the opinion of the investigator, if the patient has significant medical or psychosocial problems or unstable disease status
* Pregnant or lactating females
* Known hypersensitivity to mycophenolic acid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To test whether the addition of Myfortic improves the efficacy of prednisone plus cyclosporine for treatment of newly diagnosed chronic GvHD, as defined by the proportion of patients with efficacy success at 1 year after enrollment. | 1 year

SECONDARY OUTCOMES:
The hazard rates of efficacy success between the two arms. Loss of donor chimerism or recurrent malignancy before secondary systemic therapy and before discontinuation of all immunosuppressive meds will be treated as competing risks. | 1 year
efficacy failure, and treatment failure defined as efficacy failure or premature discontinuation of study-drug administration due to toxicity | 1 year
survival without recurrent malignancy | 1 year
Overall survival | 1 year
cumulative incidence of secondary systemic treatment for cGvHD before recurrent malignancy | 1 year
the cumulative incidence of death without recurrent or malignancy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Socié, Study Chair — Hôptial St Louis, Paris
Locations (8):
- Hopital St. Louis, Paris, France
- University Regensburg, Regensburg, Germany
- Ospedale San Martino, Genova, Italy
- University Hospital, Maastricht, Netherlands
- Hospital Clínico Universitario, Valencia, Spain
- Karolinska University Hospital, Huddinge, Sweden
- University Hospital, Basel, Switzerland
- University Faculty of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: sponsor's website — http://ebmt.org